CLINICAL TRIAL: NCT04600336
Title: A Randomized, Double-Blind, Placebo-Controlled Phase II Study of Oxybutynin Versus Placebo for the Treatment of Hot Flashes in Men Receiving Androgen Deprivation Therapy
Brief Title: Testing the Effects of Oxybutynin for the Treatment of Hot Flashes in Men Receiving Hormone Therapy for Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: A222001; UG1CA189823 (NIH); NCI-2020-07169 (Registry Identifier: NCI Clinical Trial Reporting Program)
Record Dates: First submitted 2020-10-19; First posted 2020-10-23 (Actual); Results first posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — oxybutynin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- low-dose oxybutynin (Experimental): Patients receive low-dose oxybutynin chloride (2.5 mL twice daily) PO BID on days 8-49 (6 weeks) in the absence of unacceptable toxicity.
  Interventions: Drug: Oxybutynin Chloride; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- high-dose oxybutynin chloride (Experimental): Patients receive high-dose oxybutynin chloride (5.0 mL twice daily) PO BID on days 8-49 (6 weeks) in the absence of unacceptable toxicity.
  Interventions: Drug: Oxybutynin Chloride; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- low-dose placebo (Placebo Comparator): Patients receive a low-dose placebo (2.5 mL twice daily) PO BID on days 8-49 (6 weeks). After 6 weeks, patients may cross over to experimental arm - low-dose oxybutynin per physician discretion.
  Interventions: Drug: Placebo Administration; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- high-dose placebo (Placebo Comparator): Patients receive a high-dose placebo (5.0 mL twice daily) PO BID on days 8-49 (6 weeks). After 6 weeks, patients may cross over to experimental arm - high-dose oxybutynin chloride per physician discretion.
  Interventions: Drug: Placebo Administration; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Oxybutynin Chloride — Given PO
  Arms: high-dose oxybutynin chloride; low-dose oxybutynin
Drug: Placebo Administration — Given PO
  Arms: high-dose placebo; low-dose placebo
Other: Quality-of-Life Assessment — Ancillary studies
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial compares the effect of oxybutynin versus placebo for reducing hot flashes in men receiving androgen deprivation (hormone) therapy for the treatment of prostate cancer . Androgen deprivation therapy decreases testosterone and other androgens through medications or surgical removal of the testicles. Relative to placebo, low- or high-dose oxybutynin may reduce hot flashes in men receiving androgen deprivation therapy.

DETAILED DESCRIPTION:
The primary and secondary objectives of the study:

PRIMARY OBJECTIVE:

I. To assess the effects of two doses of oxybutynin chloride (oxybutynin) on hot flash scores relative to placebo.

SECONDARY OBJECTIVES:

I. To assess study accrual rates and compliance with the therapy. II. To characterize the safety and adverse event profile of two doses of oxybutynin in the study population.

III. To evaluate the consistency of the results across the various methods used to evaluate the efficacy of oxybutynin (i.e., hot flash scores versus hot flash frequencies, mean differences versus 50% or greater reduction since baseline, single day versus full week to define patients' baseline hot flash scores).

IV. To compare patient-reported quality of life and hot flash interference, as measured by the Hot Flash Related Daily Interference Scale (HFRDIS), across arms.

V. To compare other changes in patient symptoms, as measured by the Symptom Experience Questionnaire, across arms.

OUTLINE: Patients are randomized to 1 of 4 arms in a 2:2:1:1 ratio according to the dynamic allocation scheme.

Experimental Arm (low dose): Patients receive low-dose oxybutynin chloride orally (PO) twice daily (BID) on days 8-49 (6 weeks) in the absence of unacceptable toxicity.

Experimental Arm (high dose): Patients receive high-dose oxybutynin chloride PO BID on days 8-49 (6 weeks) in the absence of unacceptable toxicity.

Placebo Arm (low dose): Patients receive low-dose placebo PO BID on days 8-49 (6 weeks). After 6 weeks, patients may cross over to Experimental Arm (low dose) per physician discretion.

Placebo Arm (high dose): Patients receive high-dose placebo PO BID on days 8-49 (6 weeks). After 6 weeks, patients may cross over to Experimental Arm (high dose) per physician discretion.

There will be a 6-week follow-up for the Placebo Arm patients who participate in the optional crossover phase.

ELIGIBILITY:
Inclusion Criteria:

* Men who are currently receiving androgen deprivation therapy (ADT) for the treatment of prostate cancer. ADT is defined by a history of orchiectomy, or ongoing usage of gonadotropin-releasing hormone agonists or antagonists. Men receiving abiraterone, but not enzalutamide, apalutamide, and darolutamide are eligible, as the latter three are metabolized by CYP3A4 and may affect oxybutynin serum concentrations.
* Patients must be on a stable dose of all hormone-directed therapies for at least 28 days prior to registration and must not be planning to discontinue this therapy for at least 42 days following registration. Patients receiving radiation therapy during the study period are eligible
* Eligible patient must have bothersome hot flashes for >= 14 days prior to registration, defined by an occurrence of >= 28 times per week and of sufficient severity to cause the patient to seek therapeutic intervention
* Life expectancy of greater than 6 months
* Eastern Cooperative Oncology Group (ECOG) performance status - 0, 1, or 2
* In order to complete the mandatory patient-completed measures, participants must be able to speak and/or read English

Exclusion Criteria:

* No current use or future planned use of any of the following agents during the study period: drugs that are not Food and Drug Administration (FDA) approved for use in humans, androgens, estrogens, progesterone analogs, gabapentin, selective serotonin reuptake inhibitor (SSRI)/serotonin and norepinephrine reuptake inhibitor (SNRI) anti-depressants, cholinergic agonists, cholinesterase inhibitors, or complementary/alternative medicine taken for the purpose of managing hot flashes. Prior use of these agents is permitted as long as they are discontinued before registration
* No current or prior use of oxybutynin
* Patients with a history of any of the following contraindications to oxybutynin are not eligible: gastroparesis or gastrointestinal obstructive disorders; significant gastric reflux symptoms not controlled by medication; ulcerative colitis; narrow-angle glaucoma; urinary retention requiring indwelling or intermittent self-catheterization within the prior 6 months; hypersensitivity to oxybutynin or any other components of the product; current uncontrolled hyperthyroidism; uncontrolled coronary artery disease or a history of myocardial infarction within the prior 12 months; New York Heart Association (NYHA) class II-IV congestive heart failure; symptomatic cardiac arrhythmias; current uncontrolled hypertension; myasthenia gravis; or dementia

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2021-10-28 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bradley J. Stish, MD, Study Chair — Mayo Clinic
Locations (103):
- United States (103):
  - Arizona Breast Cancer Specialists-Gilbert, Gilbert, Arizona
  - Arizona Center for Cancer Care-Peoria, Peoria, Arizona
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Arizona Breast Cancer Specialists-Phoenix, Phoenix, Arizona
  - Arizona Breast Cancer Specialists, Scottsdale, Arizona
  - Arizona Breast Cancer Specialists-Scottsdale, Scottsdale, Arizona
  - Arizona Center for Cancer Care-Surprise, Surprise, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - Fremont - Rideout Cancer Center, Marysville, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - Grand Valley Oncology, Grand Junction, Colorado
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Genesee Cancer and Blood Disease Treatment Center, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Ascension Saint Joseph Hospital, Tawas City, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - MU Health - University Hospital/Ellis Fischel Cancer Center, Columbia, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Nebraska Cancer Specialists/Oncology Hematology West PC - MECC, Omaha, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - AtlantiCare Health Park-Cape May Court House, Cape May Court House, New Jersey
  - AtlantiCare Surgery Center, Egg Harbor, New Jersey
  - NYP/Weill Cornell Medical Center, New York, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Messino Cancer Centers, Asheville, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Sovah Health Martinsville, Martinsville, Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Ascension Saint Elizabeth Hospital, Appleton, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Elmbrook Campus, Brookfield, Wisconsin
  - Ascension Calumet Hospital, Chilton, Wisconsin
  - Ascension Saint Francis - Reiman Cancer Center, Franklin, Wisconsin
  - Ascension Columbia Saint Mary's Hospital Ozaukee, Mequon, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Saint Joseph Campus, Milwaukee, Wisconsin
  - Ascension Columbia Saint Mary's Hospital - Milwaukee, Milwaukee, Wisconsin
  - Zablocki Veterans Administration Medical Center, Milwaukee, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Ascension Mercy Hospital, Oshkosh, Wisconsin
  - Ascension All Saints Hospital, Racine, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Ascension Medical Group Southeast Wisconsin - Mayfair Road, Wauwatosa, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The placebo arms will be half the size as the oxybutynin arms, as they will be combined to have a placebo group with the same number of patients as the two different treatment groups. This allows all patients to be blinded as to whether they are receiving active drug or a placebo. Patients randomized to the two placebo arms will be combined to form a single placebo arm for analysis.
Period: Initial Treatment
Arm/Group | Low-dose Oxybutynin | High-dose Oxybutynin Chloride | Low-dose Placebo | High-dose Placebo
Started | 28 | 28 | 15 | 11
Completed | 27 | 24 | 14 | 11
Not Completed | 1 | 4 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 0 | 0
Not completed — Adverse Event | 0 | 2 | 0 | 0
Not completed — Other complicating disease | 0 | 0 | 1 | 0
Period: Crossover Treatment
Arm/Group | Low-dose Oxybutynin | High-dose Oxybutynin Chloride | Low-dose Placebo | High-dose Placebo
Started | 0 | 0 | 11 | 8
Completed | 0 | 0 | 8 | 6
Not Completed | 0 | 0 | 3 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: All patients that were eligible and began treatment were included
Groups:
- Low-dose Oxybutynin: Patients receive low-dose oxybutynin chloride (2.5 mL twice daily) PO BID on days 8-49 (6 weeks) in the absence of unacceptable toxicity.>
  > Oxybutynin Chloride: Given PO>
  > Quality-of-Life Assessment: Ancillary studies>
  > Questionnaire Administration: Ancillary studies
- High-dose Oxybutynin Chloride: Patients receive high-dose oxybutynin chloride (5.0 mL twice daily) PO BID on days 8-49 (6 weeks) in the absence of unacceptable toxicity.>
  > Oxybutynin Chloride: Given PO>
  > Quality-of-Life Assessment: Ancillary studies>
  > Questionnaire Administration: Ancillary studies
- Placebo: Patients receive a low-dose or high-dose placebo (2.5 or 5.0 mL twice daily) PO BID on days 8-49 (6 weeks). After 6 weeks, patients may cross over to experimental arm - low-dose or high-dose oxybutynin per physician discretion.>
  > Placebo Administration: Given PO>
  > Quality-of-Life Assessment: Ancillary studies>
  > Questionnaire Administration: Ancillary studies
- Total: Total of all reporting groups
Arm/Group | Low-dose Oxybutynin | High-dose Oxybutynin Chloride | Placebo | Total
Number analyzed (Participants) | 28 | 28 | 25 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.7 (7.3) | 68.9 (7.6) | 68.8 (5.8) | 68.5 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 28 | 28 | 25 | 81
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 2
  Not Hispanic or Latino | 27 | 27 | 24 | 78
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 6 | 2 | 11
  White | 25 | 21 | 22 | 68
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 28 | 28 | 25 | 81
Daily hot flash frequency at baseline [Count of Participants; unit: Participants]
  10 or more hot flashes per day | 17 | 16 | 13 | 46
  4 to 9 hot flashes per day | 11 | 12 | 12 | 35
Hot flash duration at baseline [Count of Participants; unit: Participants]
  9 or more months | 12 | 13 | 10 | 35
  less that 9 months | 16 | 15 | 15 | 46
Number or prior hot flash therapies [Count of Participants; unit: Participants]
  0 | 22 | 20 | 19 | 61
  1 or more | 6 | 8 | 6 | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Weekly Patient-reported Hot Flash Scores
Description: Using patients' hot flash diaries, daily hot flash scores will be determined by multiplying the frequency of each defined hot flash grade (mild=1, moderate=2, severe=3, very severe=4) by the severity and summing the values over a 24-hour period. Weekly hot flash scores will be computed by averaging these hot flash scores across 7 days. A score of 0 would mean the patient experienced no hot flashes during the week, and every unit increase reflects more or more severe hot flashes experienced. A mixed model will be estimated that includes baseline and weekly hot flash scores across the 6-week treatment period. Estimates from the mixed model will be used to construct 90% confidence intervals for mean differences in hot flash score reduction from baseline to 6 weeks between the oxybutynin and placebo arms. Contrasts estimated via the mixed model will involve a two-sided t-test with alpha = .10.
Time Frame: 6 weeks post-randomization
Population: Patients that began treatment and were eligible were included in analysis
Measure: Mean (90% Confidence Interval); unit: units on a scale
Groups:
- Low-dose Oxybutynin: Patients receive low-dose oxybutynin chloride (2.5 mL twice daily) PO BID on days 8-49 (6 weeks) in the absence of unacceptable toxicity.
  >
  > Oxybutynin Chloride: Given PO
  >
  > Quality-of-Life Assessment: Ancillary studies
  >
  > Questionnaire Administration: Ancillary studies
- High-dose Oxybutynin Chloride: Patients receive high-dose oxybutynin chloride (5.0 mL twice daily) PO BID on days 8-49 (6 weeks) in the absence of unacceptable toxicity.
  >
  > Oxybutynin Chloride: Given PO
  >
  > Quality-of-Life Assessment: Ancillary studies
  >
  > Questionnaire Administration: Ancillary studies
- Placebo: Patients receive a low-dose or high-dose placebo (2.5 or 5.0 mL twice daily) PO BID on days 8-49 (6 weeks). After 6 weeks, patients may cross over to experimental arm - low-dose or high-dose oxybutynin per physician discretion.
  >
  > Placebo Administration: Given PO
  >
  > Quality-of-Life Assessment: Ancillary studies
  >
  > Questionnaire Administration: Ancillary studies
Arm/Group | Low-dose Oxybutynin | High-dose Oxybutynin Chloride | Placebo
Number analyzed (Participants) | 28 | 28 | 25
units on a scale | -9.94 [-13.10 to -6.77] | -13.95 [-17.18 to -10.73] | -4.85 [-8.20 to -1.50]
Statistical Analysis 1: Comparison: High-dose Oxybutynin Chloride vs Placebo; Test type: Superiority; p = 0.0019, t-test, 2 sided; Mean Difference (Final Values) = -9.11, 90% CI 2-sided [-13.76 to -4.46]
Statistical Analysis 2: Comparison: Low-dose Oxybutynin vs Placebo; Test type: Superiority; p = 0.0732, t-test, 2 sided; Mean Difference (Final Values) = -5.09, 90% CI 2-sided [-9.70 to -0.48]

2. Secondary Outcome: Change in Patient-reported Hot Flash Frequency
Description: Weekly hot flash frequencies will be determined by patients' hot flash diaries. A mixed model will be estimated that includes baseline and weekly hot flash frequencies across the 6-week treatment period. The mixed model and subsequent contrasts will account for the observed distribution of weekly hot flash frequencies.
Time Frame: 6 weeks post-randomization
Population: Patients that began treatment and were eligible were included in analysis.
Measure: Mean (90% Confidence Interval); unit: change in hot flashes per day
Arm/Group | Low-dose Oxybutynin | High-dose Oxybutynin Chloride | Placebo
Number analyzed (Participants) | 28 | 28 | 25
change in hot flashes per day | -4.77 [-6.05 to -3.49] | -6.89 [-8.19 to -5.58] | -2.15 [-3.50 to -0.79]

3. Secondary Outcome: Number of Patients That Experienced a Grade 3+ Adverse Event
Description: Grade 3 or higher adverse events will be assessed by the National Cancer Institute's Common Terminology Criteria for Adverse Events, version 5.0 and summarized by arm.
Time Frame: 12 weeks post-randomization
Population: Patients that began treatment were included in analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Low-dose Oxybutynin | High-dose Oxybutynin Chloride | Placebo
Number analyzed (Participants) | 28 | 28 | 26
Participants | 2 | 1 | 2

4. Secondary Outcome: Patient-reported Symptoms
Description: Patient-reported symptoms will be assessed by the Symptom Experience Questionnaire. A mixed model will be estimated that includes baseline and weekly patient-reported symptoms across the 6-week treatment period. The mean change in answers from baseline to week 6 to the item "How Distressing Was Your Experience With Hot Flashes" will be reported. Answers are given on a scale from 0 to 10 with higher scores being worse; therefore a positive number indicates a worse experience at week 6.
Time Frame: 6 weeks post-randomization
Population: Patients that began treatment, were eligible, and completed their 6 week PRO questionnaire were included in analysis
Measure: Mean (Standard Deviation); unit: average change score from baseline
Arm/Group | Low-dose Oxybutynin | High-dose Oxybutynin Chloride | Placebo
Number analyzed (Participants) | 27 | 24 | 23
average change score from baseline | -1.8 (2.74) | -3.0 (2.68) | -0.5 (2.61)
Statistical Analysis 1: Comparison: Low-dose Oxybutynin vs High-dose Oxybutynin Chloride vs Placebo; Test type: Superiority; p = 0.0120, Kruskal-Wallis

5. Secondary Outcome: Patient Accrual
Description: The time required to accrue 87 patients will be reported.
Time Frame: 26 months
Measure: Number; unit: months
Groups:
- Study: Any arm
Arm/Group | Study
Number analyzed (Participants) | 87
months | 26

6. Secondary Outcome: Patients That Completed Treatment
Description: Treatment adherence rates will be calculated by dividing the number of patients who completed treatment per protocol by the number of patients who started treatment. Treatment adherence rates will be summarized by arm.
Time Frame: 4 months
Population: All patients that began treatment and were eligible were included in analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Low-dose Oxybutynin | High-dose Oxybutynin Chloride | Placebo
Number analyzed (Participants) | 28 | 28 | 25
Participants | 27 | 24 | 25

7. Secondary Outcome: Patient-reported Hot Flash Interference
Description: A mixed model will be estimated that includes patients' scores on the Hot Flash Related Daily Interference Scale (HFRDIS) across the 6-week treatment period. The mean change in answers from baseline to week 6 to the item "Overall Quality of Life" will be reported. Answers are given on a scale from 0 to 10 with higher scores being worse; therefore a positive number indicates a worse experience at week 6.
Time Frame: 6 weeks post-randomization
Population: Patients that began treatment, were eligible, and completed their 6 week HFRDIS questionnaire.
Measure: Mean (Standard Deviation); unit: average change score from baseline
Arm/Group | Low-dose Oxybutynin | High-dose Oxybutynin Chloride | Placebo
Number analyzed (Participants) | 28 | 28 | 25
average change score from baseline | -1.0 (2.88) | -2.4 (1.89) | 0.0 (2.70)
Statistical Analysis 1: Comparison: Low-dose Oxybutynin vs High-dose Oxybutynin Chloride vs Placebo; Test type: Superiority; p = 0.0057, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: 4 months
Groups:
- Low-dose Oxybutynin - Initial Treatment: 2.5mL oxybutynin
- High-dose Oxybutynin Chloride - Initial Treatment: 5.0mL oxybutynin
- Low-dose Placebo: 2.5mL placebo
- High-dose Placebo: 5.0mL placebo
- Low-dose Oxybutynin - Crossover Treatment: 2.5mL oxybutynin - crossover treatment
- High-dose Oxybutynin Chloride - Crossover Treatment: 5.0mL oxybutynin - crossover treatment
Arm/Group | Low-dose Oxybutynin - Initial Treatment | High-dose Oxybutynin Chloride - Initial Treatment | Low-dose Placebo | High-dose Placebo | Low-dose Oxybutynin - Crossover Treatment | High-dose Oxybutynin Chloride - Crossover Treatment
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28 | 0/15 | 0/11 | 0/11 | 0/8
Serious Adverse Events (participants affected / at risk) | 2/28 | 1/28 | 0/15 | 0/11 | 1/11 | 0/8
Other Adverse Events (participants affected / at risk) | 17/28 | 23/28 | 1/15 | 4/11 | 5/11 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low-dose Oxybutynin - Initial Treatment (N=28) | High-dose Oxybutynin Chloride - Initial Treatment (N=28) | Low-dose Placebo (N=15) | High-dose Placebo (N=11) | Low-dose Oxybutynin - Crossover Treatment (N=11) | High-dose Oxybutynin Chloride - Crossover Treatment (N=8)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low-dose Oxybutynin - Initial Treatment (N=28) | High-dose Oxybutynin Chloride - Initial Treatment (N=28) | Low-dose Placebo (N=15) | High-dose Placebo (N=11) | Low-dose Oxybutynin - Crossover Treatment (N=11) | High-dose Oxybutynin Chloride - Crossover Treatment (N=8)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 4 (15) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 1 (2) | 6 (9) | 1 (1) | 0 (0) | 3 (13) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Watering eyes (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Belching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (5) | 2 (5) | 0 (0) | 0 (0) | 3 (13) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 4 (12) | 3 (9) | 0 (0) | 0 (0) | 2 (7) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 10 (34) | 18 (56) | 0 (0) | 1 (1) | 5 (14) | 4 (9)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (2) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 8 (20) | 2 (8) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Oral dysesthesia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 0 (0)
Proctitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 5 (12) | 3 (10) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (8) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (11) | 0 (0)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (12) | 0 (0)
Concentration impairment (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 5 (21) | 4 (9) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 5 (14) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (5) | 0 (0)
Insomnia (Psychiatric disorders) | 4 (14) | 2 (6) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Dysuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 2 (4) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 4 (13) | 3 (8) | 0 (0) | 0 (0) | 1 (11) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 2 (7) | 4 (10) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 4 (5) | 4 (9) | 1 (3) | 0 (0) | 1 (10) | 0 (0)
Urinary urgency (Renal and urinary disorders) | 2 (9) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urine discoloration (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (8) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hot flashes (Vascular disorders) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-14): https://cdn.clinicaltrials.gov/large-docs/36/NCT04600336/Prot_SAP_000.pdf